CLINICAL TRIAL: NCT07099014
Title: Inhaled Isoflurane for Sedation of Invasively Ventilated Patients With Cardiogenic Shock on Extracorporeal Membrane Oxygenation
Acronym: INSEPTION
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP230844; 2023-510261-94-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-16; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-06

CONDITIONS: Cardiogenic Shock, ECMO
Keywords: Cardiogenic shock, ECMO
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Propofol; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled ISOFLURANE (Experimental): Initial rate of 3 mL/h given for up to 14 days or until extubation
  Interventions: Drug: Inahled Isoflurane
- Propofol +/- Midazolam (Active Comparator): Propofol final dose 4 mg/kg/h +/- Midazolam, maximal dose 0,2 mg/kg/h
  Interventions: Drug: Propofol, midazolam

INTERVENTIONS:
Drug: Inahled Isoflurane — treatment administration
  Arms: Inhaled ISOFLURANE
Drug: Propofol, midazolam — treatment administration
  Arms: Propofol +/- Midazolam

SUMMARY:
Midazolam and propofol are the most used intravenous (IV) sedative agents, but their use is associated with well-known adverse effects such as accumulation, myotoxicity, tachyphylaxis, and unpredictable wake-up time.

For benzodiazepines, an increased tolerance, possible accumulation after long-term use, and an increased risk of acute withdrawal syndrome are reported. In patients on extracorporeal membrane oxygenation (ECMO) for cardiogenic shock, the negative hemodynamic effects of these drugs are a particular matter of concern. Besides the extracorporeal circuit itself may affect the pharmacokinetics of these IV sedatives. Indeed, drug sequestration in ECMO circuits is a well-known phenomenon influenced by drug chemo-physical properties. Given the large surface area of tubing and membrane, considerable quantities of drugs used in ECMO patients may be sequestered over a period, resulting in a significant increase in their volume of distribution. Similarly, frequent hemodilution and organ dysfunction would also contribute to an increase in the volume of distribution.

Propofol, which is lipophilic is significantly sequestrated in the circuit. Consequently, it is commonly observed that patients receiving ECMO have substantially higher sedative and analgesic drug requirements than patients without ECMO.

To date, there is no ideal concept for analgesia and sedation of patients on ECMO in the ICU.

A drug that sedates effectively but with minimal residual sedation after the end of the administration and without the aforementioned drawbacks of the current agents would be valuable.

Interestingly, a recent randomized controlled non-inferiority trial that randomized 338 patients showed that, compared with propofol, sedation with inhaled anaesthetics was non-inferior. Sedation with inhaled anaesthetics resulted in a higher rate of spontaneous breathing and a shorter wake-up time after 48h of sedation. Indeed, inhaled sedation, which has been associated with reduced opioid consumption and less delirium in ICU patients, is a promising alternative to IV sedation. Moreover, inhaled anaesthetics might be associated with less myocardial injury and lower doses of inotropic support in patients undergoing cardiac surgery. However, to date, the experience with volatile agents remains limited in patients on ECMO.

We hypothesized that the use of inhaled isoflurane with the Sedaconda anaesthetics conserving device (ACD) in cardiogenic shock patients on ECMO will reduce the mortality and increase the number of ventilation-free days at day 28 following ECMO onset compared to usual IV sedation by propofol and/or midazolam.

ELIGIBILITY:
Inclusion Criteria:

1. Cardiogenic shock on VA ECMO support for less than 24 hours
2. Patients on invasive mechanical ventilation receiving propofol and/or midazolam at the time of randomization
3. Invasive mechanical ventilation for less than 48 hours
4. Expected invasive ventilation and sedation for at least 24h, with a prescribed Richmond agitation scale target within the range of -1 to - 4
5. Social security registration (AME excluded)

Exclusion Criteria:

1. Age <18 and >75
2. Pregnancy or breastfeeding
3. Initiation of ECMO >24 hours
4. Initiation of mechanical ventilation >48 hours
5. Cardiopulmonary Resuscitation >20 minutes before randomization
6. Patient moribund on the day of randomization, SAPS II >90
7. Suspected or proven intracranial hypertension
8. Corrected QT interval > 450ms or with a known or suspected genetic predisposition to malignant hyperthermia
9. Chronic liver disease defined as a Child-Pugh score of 12-15
10. Patients ventilated with a tidal volume < 4ml/kg predicted body weight
11. Participation in another interventional study or being in the exclusion period at the end of a previous study.
12. Contraindication or allergies to isoflurane, propofol, midazolam or other halogenated anaesthetics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-10-13 (Estimated); Study Completion 2029-04-13 (Estimated)

PRIMARY OUTCOMES:
A composite hierarchical outcome composed of two components: 1) mortality, 2) number of days alive without invasive mechanical ventilation within 28 days following ECMO initiation | Day 28
  * Each patient will be compared with every other patient in the study and assigned a score (tie: 0, win: +1, loss: -1) for each pairwise comparison based on whom fared better.
  * If one patient survived on day 28 and the other did not, scores of +1 and -1 will be assigned, respectively, for that pairwise comparison. If both patients in the pairwise comparison survived at day 28, the assigned score will depend on which patient had more days free from mechanical ventilation: the patient with more ventilator-free days alive at day 28 will receive a score of +1, while the patient with fewer days will receive a score of -1. If both patients survived and had the same number of ventilator-free days on day 28, and if both patients died, they will be both assigned a score of 0 for that pairwise comparison. For each patient, scores for all pairwise comparisons will be summed, resulting in a cumulative score.

SECONDARY OUTCOMES:
Overall survival | Day 28
Number of ECMO-free days | Day 14, Day 28
Number of inotropes-free days | Day 14, Day 28
Number of ICU-free days | Day 28
Number of ventilation-free days | Day 14, Day 28
incidence of delirium | Day 28
Opioids daily consumption during invasive mechanical ventilation | Day 14
Consumption of propofol | Day 14
  consumption during invasive mechanical ventilation
Consumption of midazolam | Day 14
  consumption during invasive mechanical ventilation
Consumption of Clonidine | Day 14
  consumption during invasive mechanical ventilation
Consumption of Haloperidol | Day 14
  consumption during invasive mechanical ventilation
Consumption of dexmedetomidine | Day 14
  consumption during invasive mechanical ventilation
Incidence of drugs side effects (refractory hypertension, malignant hyperthermia) | From randomization to Day 28
  assess the safety of prolonged isoflurane inhalation during ECMO
Number of participants requiring ventricular assist device | Day 28
Number of participants undergoing heart transplantation | Day 28
Rate of side effects possibly linked to ineffective sedation (self-extubation, accidental ECMO decannulation, catheter withdrawal) | From randomization to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu SCHMIDT, MD, Study Director — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal

REFERENCES:
- [Background] Meiser A, Volk T, Wallenborn J, Guenther U, Becher T, Bracht H, Schwarzkopf K, Knafelj R, Faltlhauser A, Thal SC, Soukup J, Kellner P, Druner M, Vogelsang H, Bellgardt M, Sackey P; Sedaconda study group. Inhaled isoflurane via the anaesthetic conserving device versus propofol for sedation of invasively ventilated patients in intensive care units in Germany and Slovenia: an open-label, phase 3, randomised controlled, non-inferiority trial. Lancet Respir Med. 2021 Nov;9(11):1231-1240. doi: 10.1016/S2213-2600(21)00323-4. Epub 2021 Aug 26. PMID 34454654